CLINICAL TRIAL: NCT00104585
Title: Genetic Epidemiology of Parkinson's Disease
Brief Title: Consortium On Risk for Early-onset Parkinson's Disease (CORE PD)
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAA5609; R01NS036630 (NIH)
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; gene; environment; early-onset Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young onset Parkinson's disease: People with young onset Parkinson's disease and their family members

SUMMARY:
The purpose of this study is to investigate genetic and environmental risk factors that increase susceptibility to the development of early-onset Parkinson's disease (developed at or before age 50).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common, neurodegenerative condition. Although mostly a late-onset disorder, 10 percent of people with PD are reported to develop symptoms before the age of 50. To date, six genes have been found to be associated with PD, however the majority have been found in rare PD 'families'. Some studies have also identified a number of environmental risk factors, such as pesticide use, that appear to increase the risk of PD.

In a previous study, Dr. Karen Marder and her research team found that close family members of people with both early- and late-onset PD have a three-fold increased risk of PD compared to close family members of people without PD.

The purpose of the Consortium On Risk for Early-onset Parkinson's Disease (CORE PD) study is to identify the genetic factors that contribute to the development of early-onset Parkinson's disease, and to understand how these genetic factors interact with other genes and the environment to cause PD.

Participation in the study involves a blood draw (to look for genetic factors associated with PD), questionnaires collecting information on family and medical history, and a neurological examination. In addition participants may be contacted in the future and asked to participate in a more detailed interview. At that time, study investigators will also ask participants for permission to contact family members to invite them to participate in the study.

This research study requires participants to sign a consent form, which states that the research is voluntary and confidential. In addition, since this is a research study, genetic results are not released to participants or their family members now or in the future.

Scientists hope this multi-center study will increase the current knowledge of PD and that the identification of factors that cause PD will lead to better diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any person with Parkinson's disease in the United States
* Symptoms occurred before the age of 50
* Diagnosed by a neurologist.

Exclusion Criteria:

* Children who are <18 years of age
* Any probands who are cognitively impaired

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young onset Parkinson's disease patients
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2004-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Marder, M.D., M.PH., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States